CLINICAL TRIAL: NCT05032274
Title: Effect of Home-based Exercise Program on Visual Reliance, Cervical Spine Proprioception, and Postural Stability in Older Adults With Forward Head Posture
Brief Title: Effect of Postural Realignment on Postural Stability and Visual Reliance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5210004
Record Dates: First submitted 2021-08-16; First posted 2021-09-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Forward Head Posture
Keywords: Forward head posture; Balance; Home exercise program

STUDY DESIGN:
Intervention Model Description: single group pretest-posttest design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): The study will include one group and each participant will perform home-based exercise for 8-weeks.
  Interventions: Other: Home-based Exercise Program

INTERVENTIONS:
Other: Home-based Exercise Program — The exercise program will include chink tuck and shoulder retraction exercises. The chin tuck exercise will be performed in standing position. The shoulder retraction exercise includes activation and strengthening components. The activation component will be performed in standing position and strengthening component will be performed in prone position.

SUMMARY:
The purpose of this investigator-initiated study is 1) to investigate correlation between cervical spine joint position error (JPE) and postural stability in asymptomatic older adults with forward head posture (FHP), 2) to examine the effect of a home-based exercise program on visual reliance and cervical spine proprioception for postural stability in asymptomatic older adults with FHP, 3) to study the effect of immediate postural correction on cervical spine JPE and active range of motion (AROM), and 4) to determine participant post-intervention perception of changes in FHP, postural stability and effect on quality of life.

DETAILED DESCRIPTION:
This study will have a sample size of 50 older adults (males and females) aged 65-74 years old with FHP. This sample size will provide us with enough power to detect the needed effect size (medium effect size). The estimated attrition rate is 20%. The participants will be recruited from the local community through flyers, e-mails, and word of mouth. Study flyers will be delivered to physical therapy clinics, physician offices, and support groups with verbal description for further explanations. Potential participants who respond to the emails or flyers will be provided with a verbal description of the study.

The study will be conducted in the Department of Physical Therapy, Loma Linda University, Loma Linda. Hard copies will be stored in a locked file cabinet in a locked research laboratory and computer data will be stored on an encrypted computer in a locked research laboratory.

All data will be analyzed using Statistical Package for the Social Sciences (SPSS) version 27.0. For quantitative data, the investigators will use the General Linear Model (Mixed Factorial Analysis of Variance) and Correlation Analysis (Pearson's Correlation). Also, a statistician will be consulted to accurately analyze and interpret results. The alpha level will be set at 0.05.

Efforts will be made to keep participants' personal information confidential, but the investigators cannot guarantee absolute confidentiality. The investigators will use a pseudonym throughout the study for all recorded data so participant's actual name will not be used. Participants will not be identified by name in any publications describing the results of this study. Data in hard copy will be kept in a locked file cabinet in a locked office and electronic data will be password protected.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults aged 65-74 years with forward head posture (FHP)
2. Live independently
3. No use of assistive devices for ambulation
4. Have interest in correcting misaligned posture
5. Normal Physical Activity Readiness Questionnaire (PAR-Q+)

Exclusion Criteria:

1. Neurologic deficits
2. Disorders causing dizziness
3. Cervical spine surgery
4. Any falls in past six months
5. Medications causing frequent dizziness
6. Any health care for neck, shoulder, or low back pain past 12 months
7. Greater than minimal neck pain as determined by the Visual Analogue Scale (VAS) > 3/10
8. Neck Disability Index (NDI) > 15%
9. Forward Head Angle (FHA) < 46 degrees
10. Forward Shoulder Angle (FSA) < 52 degrees

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Change in Cervical Joint Position Error (JPE) | JPE will be measured twice (pre vs post-intervention) and each time will take approximately 25-30 minutes.
  Ability to relocate one's head and neck to pre-determined neutral position recorded in degrees.
Change in Active Cervical Spine Range of Motion (AROM) | AROM will be measured twice (pre vs post-intervention) and each time will take approximately 5 minutes
  Ability to actively move cervical spine in all six directions (flexion, extension, right and left rotation, right and left Lateral flexion). Cervical AROM will be measured in degrees.
Change in Postural Stability | Postural stability will be measured twice (pre vs post-intervention) and each time will take approximately 25 minutes
  Ability to keep center of gravity within base of support under six different testing conditions and will be scored from 0-100 by the computer software. Higher scores indicate better postural stability.
Change in Forward Head Angle (FHA) | FHA will be measured twice (pre vs post-intervention) and each time will take approximately 13 minutes.
  FHA is the angle formed between a line extending from the tragus to C7 and a vertical axis at C7. FHA will be measured in degrees.
Change in Forward Shoulder Angle (FSA) | FSA will be measured twice (pre vs post-intervention) and each time will take approximately 13 minutes.
  FSA is the angle between a line extending from C7 to acromion and the vertical axis at C7. FSA will be measured in degrees.
Post-Intervention Structured Interview | 20-25 minutes
  Post-intervention structured interview will be conducted using open-ended questions. Interviews will be recorded and transcribed verbatim. Transcriptions will be individually coded, and then group coded using qualitative research software.

SECONDARY OUTCOMES:
Change in Balance Confidence | ABC-6 will be conducted twice (pre vs post-intervention) and each time will take approximately 5 minutes.
  Subjective confidence in performing functional activities without losing balance. Activities-Specific Balance Confidence (ABC-6) scale will be used to measure balance confidence. ABC-6 scale ranges from 0 to 100 where 0 represents "no confidence" and 100 represents "complete confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Eric G Johnson, DSc, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Franz JR, Francis CA, Allen MS, O'Connor SM, Thelen DG. Advanced age brings a greater reliance on visual feedback to maintain balance during walking. Hum Mov Sci. 2015 Apr;40:381-92. doi: 10.1016/j.humov.2015.01.012. Epub 2015 Feb 14. PMID 25687664
- [Background] Sheikhhoseini R, Shahrbanian S, Sayyadi P, O'Sullivan K. Effectiveness of Therapeutic Exercise on Forward Head Posture: A Systematic Review and Meta-analysis. J Manipulative Physiol Ther. 2018 Jul-Aug;41(6):530-539. doi: 10.1016/j.jmpt.2018.02.002. Epub 2018 Aug 11. PMID 30107937
- [Background] Lee MY, Lee HY, Yong MS. Characteristics of cervical position sense in subjects with forward head posture. J Phys Ther Sci. 2014 Nov;26(11):1741-3. doi: 10.1589/jpts.26.1741. Epub 2014 Nov 13. PMID 25435690
- [Background] Silva AG, Johnson MI. Does forward head posture affect postural control in human healthy volunteers? Gait Posture. 2013 Jun;38(2):352-3. doi: 10.1016/j.gaitpost.2012.11.014. Epub 2012 Dec 7. PMID 23219786